CLINICAL TRIAL: NCT04131608
Title: Effect of Iron Deficiency Anemia on HBA1C in Patients With Diabetic Foot Ulcer Grade (1and2)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MSSAMIR, Resident doctor at INTERNAL medicine department assiut university hospital, Assiut University
Other Study IDs: HBA1C and anemia
Record Dates: First submitted 2019-09-25; First posted 2019-10-18 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-10

CONDITIONS: Iron Deficiency Anemia; HBA1C
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic foot ulcer (1and2)with iron defic: 50 diabetic patients with diabetic foot ulcer grade (1and2) with iron deficiency anemia will be applied TO
  1. cbc
  2. ferritin
  3. HBA1C
  4. ankle brachial index by duplex
  Interventions: Diagnostic Test: CBC ,Serum ferritin ,HBA1C
- diabetic foot ulcer grade(1and2)without iron deficiency anemia: 50 patients with diabetic foot ulcer grade (1and2) without iron deficiency anemia will be applied to
  1. CBC
  2. Ferritin,
  3. HBA1C
  4. ankle brachial index by duplex
  Interventions: Diagnostic Test: CBC ,Serum ferritin ,HBA1C

INTERVENTIONS:
Diagnostic Test: CBC ,Serum ferritin ,HBA1C — Diabetic patients will be applied to CBC, HBA1C and serum ferritin
  Other Names: Ankle brachial index by duplex

SUMMARY:
Diabetic foot ulcer is the commonest cause of severe limb ischemia in diabetes mellitus And development of anemia is an additional burden to the microvascular complications of diabetes

DETAILED DESCRIPTION:
HBA1C is the predominant Hemoglobin found in HBA1 fraction and it constitutes 5% of total Hemoglobin in normal adults and up to 15%in patients with diabetes mellitus HBA1C is used to diagnose diabetes and to identify individuals that are at high risk for developing diabetes Iron deficiency anemia is one of the most prevalent form of malnutrition affect 1,62 billion people whish correspond to 24,8%of the world population Ferritin is the storage form of iron so it is found to be test for distinguishing those with iron deficiency anemia from those who are not iron deficient

ELIGIBILITY:
Inclusion Criteria:

* all diabetic patients with diabetic foot ulcer grade one and two above 18 year

Exclusion Criteria:

1. patients with anemia other than iron deficiency anemia
2. Patients on anticoagulants
3. patients with blood disease 4-patients below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with diabetic foot ulcer grade one and two with or without iron deficiency anemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Iron deficiency detected by Hemoglobin level in g/dl HBA1C level in diabetic patients | Base line
  The influence of iron deficiency anemia on HBA1C in diabetic patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim S, Min WK, Chun S, Lee W, Park HI. Glycated albumin may be a possible alternative to hemoglobin A1c in diabetic patients with anemia. Clin Chem Lab Med. 2011 Oct;49(10):1743-7. doi: 10.1515/CCLM.2011.646. Epub 2011 Jun 17. PMID 21679130
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S62-9. doi: 10.2337/dc10-S062. No abstract available. PMID 20042775
- [Background] Kim C, Bullard KM, Herman WH, Beckles GL. Association between iron deficiency and A1C Levels among adults without diabetes in the National Health and Nutrition Examination Survey, 1999-2006. Diabetes Care. 2010 Apr;33(4):780-5. doi: 10.2337/dc09-0836. Epub 2010 Jan 12. PMID 20067959
- [Background] Wolffenbuttel BH, Herman WH, Gross JL, Dharmalingam M, Jiang HH, Hardin DS. Ethnic differences in glycemic markers in patients with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):2931-6. doi: 10.2337/dc12-2711. Epub 2013 Jun 11. PMID 23757434
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215